CLINICAL TRIAL: NCT03236636
Title: Comparison of Efficacy and Safety of Icaritin Versus Cinobufotalin in First-line Treatment of Advanced Hepatocellular Carcinoma Subjects: a Multicenter, Randomized, Double-blind, Double-dummy Phase III Clinical Trial
Brief Title: The Phase III Study of Icaritin Versus HUACHANSU PIAN in Hepatocellular Carcinoma Subjects
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Shenogen Biomedical Co., Ltd (Industry)
Collaborators: Chinese Academy of Medical Sciences (Other); NanJing PLA 81 Hospital (Other); Peking University Cancer Hospital & Institute (Other); Beijing Hospital (Other Government); Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other); Jinan Central Hospital (Other); Linyi Tumour Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Anhui Provincial Hospital (Other Government); The First Affiliated Hospital with Nanjing Medical University (Other); The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu Province, China (Other); Nanfang Hospital, Southern Medical University (Other); First People's Hospital of Foshan (Other); Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other); Hebei Medical University Fourth Hospital (Other); The First Hospital of Jilin University (Other); Haikou People's Hospital (Other); Fudan University (Other); West China Hospital (Other); Chongqing Traditional Chinese Medicine Hospital (Other); Chifeng Municipal Hospital (Other); The Affiliated Hospital of Hangzhou Normal University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Guilin Medical University, China (Other); The Third Xiangya Hospital of Central South University (Other); Yunnan Provincial Hospital of Traditional Chinese Medicine (Unknown); The Sixth People's Hospital of Shenyang (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNG1705ICR-1
Record Dates: First submitted 2017-07-26; First posted 2017-08-02 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Advanced HBV-Related Hepatocellular Carcinoma (HCC)
MeSH Terms: interventions — icaritin; SNG162

STUDY DESIGN:
Intervention Model Description: multicenter, randomized, double-blind, double-dummy, adaptive enrichment design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Icaritin (Experimental): Icaritin:600mg/time, 6 capsules/time(6×100mg/capsule), 2 times/day(30 minutes after breakfast, lunch and dinner), take orally, continuous administration until reach the standard of termination.
  Interventions: Drug: Icaritin
- HUACHANSU PIAN (Active Comparator): HUANCHANSU PIAN:Take orally 4 tablets/time(0.3g/tablet), 3 times/day(30 minutes after breakfast, lunch and dinner), continuous administration until reach the standard of termination.
  Interventions: Drug: HUACHANSU PIAN

INTERVENTIONS:
Drug: Icaritin — Icaritin：600mg/time, 6 capsules/time(6×100mg/capsule), 2 times/day(30 minutes after breakfast, lunch and dinner), take orally, continuous administration until reach the standard of termination.
  Other Names: SNG-162
  Arms: Icaritin
Drug: HUACHANSU PIAN — HUACHANSU PIAN:Take orally 4 tablets/time(0.3g/tablet), 3 times/day(30 minutes after breakfast, lunch and dinner), continuous administration until reach the standard of termination.
  Other Names: HUACHANSU PIAN（999）
  Arms: HUACHANSU PIAN

SUMMARY:
The enriched HBV-related advanced HCC patient population (composite biomarker score ≥ 2) and overall survival (OS) were compared between the two groups.

DETAILED DESCRIPTION:
The basis of enrichment design adjustment ： The latest published literature shows that the heterogeneity and immune tolerance of patients with hepatitis B virus (HBV) - related HCC are significantly correlated with a number of cytokines, including helper T cell subgroup 1 / 2 (Th1 / Th2) related factors. Moreover, the accumulated data show that the immunomodulatory effect of flavonoids including Icaritin is related to Th1 / Th2 factors. At the same time, the recent REACH2 study published in Lancet Oncology has successfully used serum alpha fetoprotein (AFP≥400) to enrich patients with advanced HCC. Based on the updated published data and our phase II clinical trial data, considering that the ongoing clinical trials are still in a blind state and no statistical analysis has been conducted, with consulting of clinical experts, regulatory agency advice, the protocol was amended and approved into adaptive enrichment design. Before unblended and SAP, the amendment protocol was prospectively pre-defined including sample size, patient population (CBS score positive), and event number for interim and final analysis. combined with the latest FDA clinical trial enrichment design guidelines (2019), several experts recommended to use the composite biomarkers, including IFN-γ , TNF - α and AFP, which may demonstrate the clinical advantages of the immunomodulation therapy with Icaritin for HBV-related advanced HCC patients in China with poor prognosis, but currently lack of treatment options.

Definition of enriched HBV-related advanced HCC patient:

Patient with serum composite biomarker score (CBS)≥2

Enrichment design amendment:

Based on our previous phase II data of Icaritin collected from HBV-related advanced HCC patients and the related literature, we assume that the mOS of the enriched population (CBS≥2) is 420 days (14 months) in the experimental group and 240 days (8 months) in the HUACHASHU control group; the HR of the experimental group relative to the control group is 0.57. A total of 106 target death events and 130 evaluable subjects were required for the enrichment. Once the amendment protocol be effective, the enriched and non-enriched patients will be continuously randomized into the experimental and the control arms accordingly (1:1). When the number of enrolled cases reaches 280, or 60% of events (64) of 106 deaths has been observed in the enriched population, interim analysis will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Only patients who meet all the following criteria are included in the study:

  1) Age≥18years, no gender restriction; 2) Advanced or metastatic HCC patients in strict compliance with the "Primary Liver Cancer Diagnosis and Treatment Standard" (2017 Edition) issued by the National Health and Family Planning Commission, clinical diagnostic criteria and/or diagnosed by pathology /cytology, patients who fail to undergo liver surgery and/or other local treatment (ablation or hepatic artery intervention), or patients who have recurrence and progression after surgery and/or other local treatment; 3) Not previously accepted first-line system therapy (systemic chemotherapy, molecular targeting, immunotherapy and research medication, etc.) for advanced or metastatic HCC, including but not limited to systematic chemotherapy with oxaliplatin, sorafenib, PD-1/PD-L1 antibody, Icaritin and cinobufotalin, etc.; 4) Liver surgery was performed more than 3 months ago, ablation or interventional treatment of hepatic artery was performed more than 4 weeks ago, and the adverse reactions returned to normal; After surgery or other local treatment, if patients have gone beyond the norm for systemic adjuvant chemotherapy, it will need more than 6 months after the chemotherapy, and disease progression and / or metastasis have occurred; 5) For patients who are not suitable for first-line treatment of advanced HCC which is recommended in "Primary Liver Cancer Diagnosis and Treatment Standard." issued by the National Health and Family Planning Commission, it's mainly due to partial blood test indicators (See the relaxed scope in 11th inclusion criteria ) or other indicators (Including mild ascites and so on) which are not suitable for the existing first-line standard treatment; Or in particular cases, the patients insist on refusing to accept the existing first-line standard treatment(For example, patients feel that their physical condition is weak and / or economic constraints, which must be strictly mastered and controlled); 6) 2 weeks before the first medication of the trial, there is no use of modern Chinese medicine preparation with liver cancer indication, including Delisheng injection, Kanglaite injection or soft capsule, Aidi injection or Considi injection, elemene injection/oral liquid, 1) 7) no use of blood transfusion or blood products, no use of hematopoietic stimulating factor, no transfusion of albumin or blood products 14 days before screening; 8) According to the evaluation criteria of solid tumor reaction (RECIST 1.1), it has at least one measurable target lesion, which defined as non-lymph node lesions with the longest diameter larger than 10mm, lymph node lesions with the short diameter larger than 15mm; the lesions previously received local treatment such as ablation or hepatic artery interventional therapy should be detected by computed tomography (CT) / magnetic resonance imaging (MRI) and according to RECIST1.1, It's sure that disease progression has occurred and the longest diameter is more than 1.0cm,it can be used as a measurable target lesions; 9) The Child-Pugh score of liver function is grade A or better grade B (score≤7); 10) The ECOG score of physical condition is 0-1; 11) Expected survival time≥12 weeks; 12) The function of the main organs is basically normal and meets the following requirements:

  ①Marrow: There is no blood transfusion and use of hematopoietic cell stimulating agent, including granulocyte colony stimulating factor (G-CSF)within 14 days before screening, platelet≥60×10E9/L, hemoglobin≥ 85g/L, white blood cell≥3.0×10E9/L; After a thorough measurement of the patient's condition, the above three items can be appropriately relaxed by the principal researchers at the research centre as: platelet 50 ~60×10E9/L, hemoglobin 80~85g/L, white blood cell 2.5 ~3.0×10E9/L (contains critical values);

  ②Liver: Total bilirubin≤1.5 times of the upper limit of normal(ULN), Aspartate aminotransferase (AST) and alanine aminotransferase (ALT)≤5 × ULN; albumin≥ 28g/L;

  ④ Kidney: Serum creatinine≤ 1.5 x ULN, or creatinine clearance rate≥ 50ml/min; 13) If HBV-DNA≥104 copies/ml(2000IU/ml), antiviral therapy must be done first, the patient can be included in the group until HBV-DNA<104 copies /ml(2000IU/ml); and continue to take antiviral drugs, monitor liver function and hepatitis B virus load; 14) Women of childbearing age must receive pregnancy tests 14 days before treatment and the results are negative; Men of childbearing age need effective contraception during treatment and within 3 months after treatment; 15) Patients are volunteered to join the study, sign the informed consent, have good compliance and cooperate with follow-up; 16) The subjects do not participate in other clinical trials within 4 weeks before screening; If the subject fails in other test screening, but meets the requirements of this test, then can be enrolled.

Exclusion Criteria:

* Patients who meet any of the following criteria are not allowed to enter the test:

  1. Imaging examination shows that HCC liver tumors are huge (≥60% of the liver volume), or cancer embolus of portal trunk (occupying ≥50% of the vascular diameter), or cancer embolus invading mesenteric vein or inferior vena cava;
  2. Middle or higher ascites which is clinically significant, it requires therapeutic abdominal paracentesis /drainage, or the Child-Pugh score > 2;
  3. Local anticancer therapy (including surgery, ablation, hepatic arterial chemotherapy, embolization or radiotherapy) or major surgery was performed 28 days prior to randomization;
  4. Hepatocholangiocarcinoma and fibrolamellar cell carcinoma; In the past 5 years or at the same time, there were other malignancies, except cervical carcinoma in situ, previously treated basal cell carcinoma and superficial bladder tumor (Ta, Tis, T1);
  5. Pregnant or lactating women;
  6. The patient suffers from CTCAE classification type II or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmia; and/or NYHA standard III to IV cardiac dysfunction.
  7. Allograft transplants including liver transplantation were performed previously, or a liver transplant was planned during the trial;
  8. Hepatic encephalopathy and / or hepatic nephropathy occurred within 6 months;
  9. Patient with active hepatitis C, that is, anti -HCV positive or HCV-RNA positive and abnormal liver function;
  10. Human immunodeficiency virus (HIV) tests are positive or severe infection requiring systemic treatment with antibiotics;
  11. Inability to swallow, chronic diarrhea or intestinal obstruction that significantly affecting medication intake and absorption;
  12. Having a history of digestive tract bleeding within 6 months, or with a clear gastrointestinal bleeding tendency, including local active ulcerative lesions, positive fecal occult blood;
  13. The patient has or is suspected to have known active autoimmune disease;
  14. If a central nervous system metastasis is known and a metastasis of the central nervous system is suspected, the cranial MRI examination should be performed to exclude it;
  15. Abnormal coagulation function: international normalized ratio (INR) >1.5 or prothrombin time (PT) >16S;
  16. There is a history of schizophrenia or psychotropic substance abuse;
  17. Known to be allergic or intolerant to Icaritin or cinobufotalin and excipients;
  18. Other conditions that researchers believe discourage patients from participating in trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2017-09-08 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 2-4 years
  OS is defined as the time from randomization to died from any cause. For the subjects who failed to visit, deletion is performed on the final date of knowing the survival of the subjects, for subjects who still survive, deletion is performed on the data expiration date.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2-3 years
  PFS is defined as the date from randomization to the first radiographic record of disease progression or death (whichever occurs first). See the Statistical Analysis Plan (SAP) for the definition of PFS deletion rule.
Time to progress（TTP） | 2-3 years
  TTP is defined as the date from randomization to the first radiographic record of disease progression, see the Statistical Analysis Plan(SAP) for the definition of TTP deletion rule.
Overall response rate (ORR) | 2-3 years
  ORR is defined as the proportion of subjects achieving optimal overall efficacy such as CR or partial remission (PR).
Overall disease control rate (DCR) | 2-3 years
  DCR is defined as the proportion of subjects achieving optimal overall efficacy such as CR, PR or stable disease (SD).
Assessment on Quality of life 1 | 2-4 years
  Quality of life (QOL) changes: Quality of life scores are assessed with EORTC QLQ-C30 and compared with baseline values.
Assessment on Quality of life 2 | 2-4 years
  Quality of life (QOL) changes: Quality of life scores are assessed with EORTCQLQ-HCC-18 and compared with baseline values.

OTHER OUTCOMES:
Biomarker analysis of proteome level (Immunohistochemical method) | 2-4 years
  Baseline expression or expression changes of programmed cell death ligand 1 (PD-L1), heterogeneous ribonucleoprotein A2/B1 (hnRNPAB1) and interleukin -6 (IL-6) and so on.
Genome level (DNA, mRNA, miRNA) biomarker analysis | 2-4 years
  Genetic variation(Liver cancer driver genes and hotspot gene mutations, such as IDH1/2, JAK2/3, PD-L1/2), expression levels of oncogenes and immune related genes(Gene copy number and RNA expression level) and epigenetics cohort analysis

CONTACTS AND LOCATIONS:
Overall Officials: Yan Sun, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Shukui Qin, Principal Investigator — NanJing PLA 81 Hospital
Locations (28):
- China (28):
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Hospital, Beijing, Beijing Municipality
  - General Hospital of Chinese Armed Police Forces, Beijing, Beijing Municipality
  - Guang'anmen Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing Traditional Chinese Medicine Hospital, Chongqing, Chongqing Municipality
  - The First People's Hospital of Foshan, Foshan, Guangdong
  - Affiliated Hospital of Guilin Medical University, Guilin, Guangxi
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Haikou People's Hospital, Haikou, Hainan
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Eastern Theater General Hospital,QinHuai District Medical Area, Nanjing, Jiangsu
  - The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu
  - The Affiliated Tumor Hospital of Nantong University, Nantong, Jiangsu
  - First Hospital of Jilin University, Changchun, Jilin
  - The Sixth People's Hospital in Shenyang, Shenyang, Liaoning
  - Chifeng Municipal Hospital, Chifeng, Neimenggu
  - Jinan Central Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Yunnan Provincial Hospital of Traditional Chinese Medicine, Kunming, Yunnan
  - The Affiliated Hospital of Hangzhou Normal University, Hangzhou, Zhejiang
  - Nanfang Hospital of Southern Medical University, Guangzhou

IPD SHARING:
Plan to Share IPD: No